CLINICAL TRIAL: NCT03534830
Title: Estimated Levator Ani Subtended Volume (eLASV): A Novel Assay for Predicting Surgical Outcomes in Pelvic Organ Prolapse
Brief Title: A Novel Assay for Predicting Surgical Outcomes in Pelvic Organ Prolapse
Acronym: eLASV
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 00031263
Record Dates: First submitted 2018-03-15; First posted 2018-05-23 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Prolapse Genital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- eLASV > 38.5: exposed group of patients with an eLASV at or above 38.5 on a pre-operative MRI.
  Interventions: Diagnostic Test: MRI
- eLASV < 38.5: non-exposed group of patients with an eLASV less than 38.5 of pre-operative MRIs
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — pre-operative MRI to be performed on all patients and then based on the imaging studies, the patient will be divided into the two comparative cohorts

SUMMARY:
The research objective of this proposal is to investigate the clinical utility and validity of eLASV as a personalized marker for women's individual risk of recurrence for pelvic organ prolapse following advanced surgical procedures. Estimated levator ani subtended volume (eLASV) is a reproducible magnetic resonance image of the female pelvis that objectively quantifies the integrity of the pelvic floor levator ani muscles. A woman's levator ani muscle anatomical shape is unique to her as a result of her own individual lifetime risk for development of pelvic floor dysfunction. The novelty of eLASV as a measurement of muscle integrity, separates it methodology from the solitary of diagnosing partial trauma or defects as previously published within the literature. eLASV measurements have the potential to identify women at increased risk for surgical failure and may be used as a prognostic tool to aid in future counseling and stratification of patients into surgical options for treatment of pelvic organ prolapse.

DETAILED DESCRIPTION:
Pelvic floor disorders affect millions of women within the United States daily, with nearly 25% of all women currently have some form of pelvic floor dysfunction [1]. An estimated 200,000 women undergo surgery annually for pelvic organ prolapse [4-6], and recent projections estimate that the number will increase to approximately 250,000 by year 2050 [7]. Up to 30% of these women, will undergo a second surgical procedure for recurrence of prolapse following their first surgery [2]. Astoundingly, resulting in 60,000 - 75,000 women a year undergoing a second advanced gynecological surgical procedure for pelvic organ prolapse consequently increasing the patients' perioperative risk and the overall cost of women's healthcare nationwide.

Levator ani muscle plays an important role in pelvic support. Weakening or direct trauma to the muscle is currently the best-defined pathogenesis for development of pelvic organ prolapse and for the recurrence of prolapse after surgical repair [7-13]. Levator ani avulsion has been demonstrated to be a clinical predictor of cystocele recurrence following anterior colporrhaphy with native tissue and with mesh augmentation [11,12]. However, further studies are warranted to investigate of levator ani muscle integrity as a predictor for surgical outcomes after more advance surgical procedures.

The investigators demonstrated an objective measure of levator ani muscle integrity (eLASV) calculated from standard 2D dynamic pelvic MRI measurements (H-line and M-line) obtained directly from radiology reports along with one 2D linear measurement that is easily obtained from radiographic images [13-15]. The novelty of eLASV as a measurement of the entire muscle integrity, separates it methodology from the solitary of diagnosing partial trauma or defects as previously published within the literature. eLASV is a novel objective measurement of levator ani muscle integrity and measures all three portions of the muscle (puborectalis, pubococcygeus, and iliococcygeus) as a whole complex. Transvaginal and transperineal ultrasonography along with CT scans or xRays of the pelvic floor are unable to image at the high level resolution imperative for complete reconstruction of the entire levator ani muscle.

Each woman's levator ani muscle anatomical shape is unique to her as a result of her own individual lifetime risk for developement of pelvic floor dysfunction. Consider the levator ani muscle as a kitchen bowl varying in different shapes and sizes for each individual woman. Now consider filling these varying shapes and sizes of the kitchen bowls with water, eLASV is the objective three dimensional measurement of the volume of water contained within each different muscle complex.

When the volume of eLASV is elevated, it represents a measurable change in the anatomical shape of the muscle as a result of loss of the muscle integrity for support of the pelvic floor. As Decreased support of the levator ani muscle within the pelvic floor will result in an increased strain on the supportive ligament structures within the female pelvis [16,17]. Increased strain on the supportive structures including the uterosacral ligament, sacrospinous ligament, paravaginal support, etc., could result in an increased risk of recurrence for prolapse following advance pelvic reconstructive surgery.

eLASV may have the potential to identify women at increased risk for surgical failure and could be used as a prognostic tool to aid in future counseling of patients on surgical options for treatment of pelvic organ prolapse. Identification of women at an increased risk for surgical failure following advanced surgical procedures would be invaluable in a surgical subspecialty that has a reoperation rate as high as 30% after a primary surgery [2].

Personalized medicine and patient selection thus far has played a very small role in the discussion regarding the use of mesh versus native tissue repair in female pelvic reconstructive surgery. Patient stratification into certain reconstructive procedures will likely change once clinicians become better at diagnosing levator ani trauma and identify patients at high risk of prolapse recurrence after reconstructive surgery [8]. Abdominally placed mesh, either via robotically, laparoscopically, or open, for a sacral colpopexy is considered the gold standard for apical suspension in patients with pelvic organ prolapse [18]. However, there is an increased concern for the use of synthetic mesh in reconstructive pelvic surgery [19].

This study represents a step in the direction of identifying patients at increased risk for surgical failure and the potential of stratifying future patients into specific surgical procedures based on their own individual likelihood of success vs failure after an advanced pelvic reconstructive procedure improving patient outcomes.

Approach: The specific aims of this project will be fulfilled through a combined qualitative and quantitative approach. The investigators plan to test the feasibility of executing a prospective cohort trial investigating the clinical utility of eLASV as a preoperative biomarker and prognostic tool to predict surgical outcomes in pelvic organ prolapse by assessing the study design/process, resources available, management and time barriers, along with the scientific merit of the study. The investigators will also plan to test the validity of eLASV calculation and pilot test eLASV as a biomarker at 38.5 to predict surgical outcomes for laparoscopic uterosacral ligament suspension. The investigators will then use the information gathered from our pilot study to refine or modify the research methodology to develop a larger, NIH grant supported prospective cohort control trial.

ELIGIBILITY:
Inclusion Criteria

* Greater than or equal to 18 years old
* English speaking
* Willing to sign an informed consent
* Stage III pelvic organ prolapse
* Undergoing uterosacral ligament suspension for pelvic organ prolapse Exclusion Criteria
* Women who do not meet the inclusion criteria.
* Inability to undergo a pelvic MRI
* Having a different apical suspension procedure for pelvic organ prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 50 women total with symptomatic stage III pelvic organ prolapse who elect to proceed with surgical intervention within the Division of Urogynecology at University of South Florida (USF) Department of Obstetrics and Gynecology.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Surgical failure after apical prolapse repair | one year
  Surgical failure will be a single composite outcome that will be defined by any of the following information: presence of anatomic bulge beyond the hymen (within any compartment: anterior, posterior, or apical), sensation of a symptomatic vaginal bulge, or the need for repeat treatment for prolapse via pessary or surgery

SECONDARY OUTCOMES:
Repeatability of measurement | one year
  Repeatability of MRI measurements to calculate eLASV
Reliability of measurement-inter observer | one year
  Inter observer reliability of measurements of 2d images to calculate eLASV
Reliability of measurement intra observer | one year
  Intra-observer reliability of measurements of 2d images to calculate eLASV

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wyman AM, Salemi JL, Lai-Yuen S, Greene KA, Bassaly R, Kedar R, Hoyte L. Estimated Levator Ani Subtended Volume: A Predictive Biomarker for Surgical Outcomes Following Native Tissue Apical Repair. Female Pelvic Med Reconstr Surg. 2022 Jun 1;28(6):385-390. doi: 10.1097/SPV.0000000000001142. Epub 2022 Mar 4. PMID 35234178